CLINICAL TRIAL: NCT00104013
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, 18-Month Study of the Efficacy of Xaliproden in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Brief Title: Study of Xaliproden (SR57746A) in Patients With Mild-to-Moderate Dementia of the Alzheimer's Type
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC2724; SR57746A
Record Dates: First submitted 2005-02-18; First posted 2005-02-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — xaliproden

INTERVENTIONS:
Drug: xaliproden (SR57746A)

SUMMARY:
The purpose of this study is to assess xaliproden's potential capacity of slowing the deterioration of cognitive and global functions in patients with mild to moderate Alzheimer's disease. The patients participating in this study will take orally once daily xaliproden or placebo (inactive substance pill).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease using NINCDS-ADRDA criteria

  * Mild to moderate degree of severity of dementia as assessed by the Mini-Mental Status Examination score of 16 to 26 (inclusive)
  * Potential participant may be treated with conventional Alzheimer's disease therapy and must be on a stable dose for at least 6 months prior to the randomization and during the entire study period
  * Potential participant must have a reliable caregiver and must be living in a community or in an assisted living facility
  * Mother tongue is English, Spanish or French (oral and written fluency)
  * Signed informed consent from potential participant or legal representative and identified caregiver

Exclusion Criteria:

* Potential participant with any other cause of dementia.
* Potential participant with serious health problems other than Alzheimer's disease
* Use of an investigational drug within two months prior to randomization or during this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1455 (Actual)
Dates: Start 2003-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease assessment scale-cognitive, clinical dementia rating sum of boxes.

SECONDARY OUTCOMES:
Mini-Mental State Examination, Alzheimer's Disease assessment scale-activities of daily life.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (41):
- United States (32):
  - Neurological Physicians of Arizona, Inc., Mesa, Arizona
  - Pivotal Research Centers, Mesa, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Northwest NeuroSpecialists, Tucson, Arizona
  - Optimum Health Services, Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - Univ. of CT Health Center, Farmington, Connecticut
  - CNS Healthcare, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - Memory Disorder Center, Pompano Beach, Florida
  - Neurological Center, Fort Wayne, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Hartford Research Group, Florence, Kentucky
  - Lexington Clinic, Lexington, Kentucky
  - LSUHSC Geriatric Psychiatry, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Synergy Medical, Saginaw, Michigan
  - University Medical Center, Dept. of Psychiatry Clinical Trials, Jackson, Mississippi
  - Radiant Research, Inc., St Louis, Missouri
  - Center For Emotional Fitness, Moorestown, New Jersey
  - Ubhc/Umdnj667, Piscataway, New Jersey
  - The Ohio State University, Columbus, Ohio
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Alzheimer's Research & Clinical Programs, North Charleston, South Carolina
  - Harmony Research, Inc, Johnson City, Tennessee
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Grayline Clinical Drug Trial, Wichita Falls, Texas
  - The Innovative Clinical Research Center, Alexandria, Virginia
  - Eastern Virginia Medical School - The Glennan Center For Geriatrics "Gerontology", Norfolk, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanfoi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com